CLINICAL TRIAL: NCT02840370
Title: Effect of Transcranial Direct Current Stimulation of the Prefrontal Cortex on Language Production in Aphasic Patients: a Multicentre Experimental Study With a Placebo-controlled and Double Blind Crossover Design
Brief Title: Effect of Stimulation of the Prefrontal Cortex on Language Production in Aphasic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jean-Marie Annoni (Other)
Collaborators: University Hospital, Geneva (Other); Hôpital Cantonal de Fribourg (Unknown)
Responsible Party: Sponsor-Investigator, Jean-Marie Annoni, Prof. Dr. med., University of Fribourg
Organization: University of Fribourg (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: SNF325130_156937_3
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Aphasia
Keywords: transcranial direct current stimulation; aphasia; language production; prefrontal cortex
MeSH Terms: conditions — Aphasia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- transcranial direct current stimulation (Experimental): tDCS
  Interventions: Device: transcranial direct current stimulation
- Sham tDCS (Sham Comparator): S-tDCS
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: transcranial direct current stimulation — In tDCS, the prefrontal cortex is stimulated during 20minutes through a weak constant electric current (1-2 mA) through two electrodes in a non-invasive and painless manner.
  Arms: transcranial direct current stimulation
Device: Sham tDCS — S-tDCS refers to a control condition in which the subject will receive a brief current in the beginning in order to induce a similar sensation on the scalp as in tDCS, and then the stimulator remains off for the rest of the stimulation time.
  Arms: Sham tDCS

SUMMARY:
The purpose of this study is to investigate whether transcranial direct current stimulation (tDCS) of the prefrontal cortex (PFC) influences lexical access and language production. The experimental paradigm will assess the impact of prefrontal stimulation by tDCS versus sham tDCS (S-tDCS) over the PFC of patients with chronic post-stroke aphasia during three language production tasks and a nonverbal executive functions task.

DETAILED DESCRIPTION:
Background:

Language processing is a complex brain function supported by a large network, including domain-specific language areas as well as domain-general cognitive-control networks (Friederici & Gierhan, 2013). Noninvasive brain stimulation, such as transcranial direct current stimulation (tDCS), is increasingly being used as a promising therapeutic tool for psychiatric and neurological diseases (Tortella et al., 2015; Flöel, 2014). In the language domain, several studies revealed that tDCS over languagespecific areas induces changes in cortical function that enhances the recovery of language abilities in patients with post-stroke aphasia (Torres, Drebing & Hamilton, 2013; Monti et al., 2013). Beneficial effects of tDCS have also been found for stimulation over more domain-general cognitive control regions. Although research on non-invasive brain stimulation and aphasia reveals promising results, studies investigating the modulation of cognitive control-networks on lexical access are rare. Given the importance of a successful interplay between prefrontal and domain-specific language areas, possible therapeutic effects of tDCS over the prefrontal cortex (PFC) in aphasia can be of high value for rehabilitation and basic research.

Procedure:

A planned total of 30 patients will be included. In a first visit, the severity of aphasia, the medical history as well as inclusion/exclusion criteria will be evaluated. After this visit, patients will undergo two tDCS sessions (one tDCS and one S-tDCS session) with a one week interval between the sessions. Each session consists of an online (during stimulation) and an offline assessment (within 30 minutes after stimulation). Three language tasks and a nonverbal executive function task will be conducted online as well as offline in each of the two sessions (tDCS and S-tDCS).

ELIGIBILITY:
Inclusion Criteria:

* Chronic aphasia due to ischemic or haemorrhagic stroke (> 6 months post-stroke)
* French as dominant language
* Right-handedness
* Left hemisphere lesion with intact bilateral PFC

Exclusion Criteria:

* Diagnosed dementia or psychiatric comorbidity
* Epileptic seizure within the last 12 months
* Metallic head implants
* Pacemaker
* Inability to understand procedures or insufficient language production abilities
* pregnancy
* strong headache on the days of the tDCS sessions
* consumption of alcohol and/or unprescribed drugs on the days of the tDCS sessions or on the day before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-05; Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Language production | up to 30 min
  Picture naming task, repetition task and verbal fluency task

SECONDARY OUTCOMES:
Nonverbal executive functions task | up to 30 min

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Annoni, Prof. Dr., Principal Investigator — University of Fribourg
Locations (3):
- Switzerland (3):
  - Laboratory for Cognitive and Neurological Sciences, Fribourg
  - Hôpital Cantonal de Fribourg, Fribourg
  - University Hospital Geneva, Geneva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friederici AD, Gierhan SM. The language network. Curr Opin Neurobiol. 2013 Apr;23(2):250-4. doi: 10.1016/j.conb.2012.10.002. Epub 2012 Nov 9. PMID 23146876
- [Background] Tortella G, Casati R, Aparicio LV, Mantovani A, Senco N, D'Urso G, Brunelin J, Guarienti F, Selingardi PM, Muszkat D, Junior Bde S, Valiengo L, Moffa AH, Simis M, Borrione L, Brunoni AR. Transcranial direct current stimulation in psychiatric disorders. World J Psychiatry. 2015 Mar 22;5(1):88-102. doi: 10.5498/wjp.v5.i1.88. PMID 25815258
- [Background] Floel A. tDCS-enhanced motor and cognitive function in neurological diseases. Neuroimage. 2014 Jan 15;85 Pt 3:934-47. doi: 10.1016/j.neuroimage.2013.05.098. Epub 2013 May 30. PMID 23727025
- [Background] Torres J, Drebing D, Hamilton R. TMS and tDCS in post-stroke aphasia: Integrating novel treatment approaches with mechanisms of plasticity. Restor Neurol Neurosci. 2013;31(4):501-15. doi: 10.3233/RNN-130314. PMID 23719561
- [Background] Monti A, Ferrucci R, Fumagalli M, Mameli F, Cogiamanian F, Ardolino G, Priori A. Transcranial direct current stimulation (tDCS) and language. J Neurol Neurosurg Psychiatry. 2013 Aug;84(8):832-42. doi: 10.1136/jnnp-2012-302825. Epub 2012 Nov 8. PMID 23138766